CLINICAL TRIAL: NCT05449145
Title: The Effects of Vitamin D Plus Omega-3 Polyunsaturated Fatty Acids in Patients With Episodic Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kuang Tien General Hospital (Other)
Responsible Party: Principal Investigator, Chun-pai Yang, MD, Chief, Department of Neurology, Kuang Tien General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KTGH11017
Record Dates: First submitted 2022-06-22; First posted 2022-07-08 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Episodic Migraine
Keywords: episodic migraine; prevention; VitD; fish oil
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): MCT oil (first 4-week) plus Omega-3 FA (second 4-week)
  Interventions: Dietary Supplement: Non-Vitamin D
- Vitamin D (Experimental): Vit D (first 4-week) plus Omega-3 FA (second 4-week)
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — 1st week: Vitamin D 82285.71 IU per day (total dose: 576000IU per week); 2th to 4th week: Vitamin D 41142.86 IU per day (total dose: 288000IU per week); 5th to 8th week: fish oil 2 capsules per day（each capsule contains EPA 900mg)
  Arms: Vitamin D
Dietary Supplement: Non-Vitamin D — 1st week: 95% MCT oil 5.71 ml per day (total dose: 40 ml per week); 2th to 4th week: 95% MCT oil 2.86 ml per day (total dose: 20 ml per week); 5th to 8th week: fish oil 2 capsules per day（each capsule contains EPA 900mg)
  Arms: Placebo

SUMMARY:
First, the aims of this study are to explore the effect of vitamin D versus placebo in the prevention of episodic migraine. Second, we would like to compare and evaluate the effect of vitamin D plus omega-3 fatty acids versus placebo plus omega-3 fatty acids in terms of migraine frequency, symptom severity, and associated complications.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of supplementing with Omega-3 fatty acids and vitamin D on the prevention of muscle atrophy and lifestyle performance in migraine patients. Furthermore, it aims to understand the biological mechanisms of action of Omega-3 fatty acids and vitamin D in decreasing migraine attacks, the severity of headaches, and associated complications, as well as inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-65 years
2. Episodic migraine diagnosis with ICHD-3
3. Baseline migraine days between 4 and 15 days per month
4. Episodic migraine without or without aura
5. Blood Vit D< 30ng/mL at baseline
6. With completed informed consent

Exclusion Criteria:

1. Non-migraine (ex: tension-type headache or secondary headache)
2. Having major head trauma in the past
3. Alcoholism within 1 year
4. Patients with abnormal liver and kidney function and patients with other serious diseases such as infection with any inflammation
5. Pregnant women or women who are still breastfeeding
6. Those who are unable to cooperate with the progress of the trial and who have participated in other clinical studies.
7. Patients with abnormal coagulation function or taking anticoagulant drugs
8. Weight < 45 kg or > 80 kg
9. Abnormal parathyroid function, intestinal dysfunction, hypercalcemia (total calcium ion concentration in blood> 2.6 mmol/L)
10. Conditions with high risk of hypercalcemia, such as: Metastatic cancer, Sarcoidosis, Multiple myeloma, Primary hyperparathyroidism
11. Those who are allergic to fish or fish oil
12. Vegetarian
13. Taking beta-blockers, antiepileptic drugs, calcium ion blockers, antidepressants or hormonal preparations in the past month
14. Using vitamin D (> 3000 IU/day), calcium tablets, estrogen drugs, bisphosphonates, and other drugs to treat bone diseases.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Change of migraine days per month from baseline | 12nd week
  From questionnaires

SECONDARY OUTCOMES:
Change of Migraine Disability Assessment (MIDAS) score from baseline | 12nd week
  Using Migraine Disability Assessment (MIDAS) score with a decreased score from baseline reflecting migraine improvement.
  1. MIDAS grade I (score 0-5) : Little or No Disability
  2. MIDAS grade II (score 6-10) : Mild Disability
  3. MIDAS grade III (score 11-20) : Moderate Disability
  4. MIDAS grade IV (score 21+) : Severe Disability
Change of Hospital Anxiety and Depression Scale (HADS) from baseline | 12nd week
  The Hospital Anxiety and Depression Scale (HADS) is a score ranging from 0 to 21 with a decreased score from baseline reflecting improvement.
  Scores of:
  1. 0-7 (Normal)
  2. 8-10 (Mild)
  3. 11-15 (Moderate)
  4. 16-21 (Severe)
Change of Visual Analogue Scale (VAS) from baseline | 12nd week
  Visual Analogue Scale (VAS) is a pain rating scale ranging from 0 to 10, and a higher score indicates greater pain. A decreased score from baseline reflecting improvement.
Change of Pittsburgh Sleep Quality Index (PSQI) from baseline | 12nd week
  Pittsburgh Sleep Quality Index (PSQI) is a score ranging from 0 to 21 with the higher total score indicating worse sleep quality. A decreased score from baseline reflecting improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Pai Yang, MD, Principal Investigator — Chief, Department of Neurology
Locations (1):
- Kuang Tien General Hospital, Taichung, Taiwan